CLINICAL TRIAL: NCT00857779
Title: A Multicentre Randomised Phase II Clinical Trial to Demonstrate Equivalent Pharmacodynamic Efficacy and Tolerability of Two Updosing Schedules for ALK-Flex SQ
Brief Title: Study on Pharmacodynamic Parameter and Tolerability With Subcutaneous Immunotherapy in Grass Pollen Allergic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AF-H-01
Record Dates: First submitted 2009-03-05; First posted 2009-03-09 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Rhinitis; Conjunctivitis; Asthma
Keywords: allergen immunotherapy; allergy to grass pollen
MeSH Terms: conditions — Rhinitis; Conjunctivitis; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- subcutaneous immunotherapy (Active Comparator): subcutaneous immunotherapy using a slow updosing schedule
  Interventions: Biological: subcutaneous immunotherapy
- subcutaneous injections (Active Comparator): subcutaneous immunotherapy using a fast updosing schedule
  Interventions: Biological: subcutaneous immunotherapy

INTERVENTIONS:
Biological: subcutaneous immunotherapy — 7 injections
  Other Names: AVANZ

SUMMARY:
The aim of this study is to test the pharmacodynamic equivalence with respect to IgE-blocking factor and to compare the tolerability of two different updosing schedules with ALK-Flex SQ

ELIGIBILITY:
Inclusion Criteria:

* A clinical history of grass pollen induced allergic rhinoconjunctivitis of two years or more requiring treatment during the grass pollen season
* Lack of adequate relief with symptomatic medication during the previous grass pollen season
* Positive Skin Prick Test (SPT) response to Phleum pratense (wheal diameter >= 3mm) currently performed or not older than 60 days before screening

Exclusion Criteria:

* FEV1 < 70% of predicted value at screening
* Bronchial asthma corresponding to GINA step 3 or more, even if controlled
* History of asthma exacerbation or emergency visit or admission for asthma in the previous 12 months
* Previous treatment by immunotherapy with grass pollen allergen or any other allergen within the previous 5 years
* Exclusion criteria in accordance with contraindications in the SPC of ALK-Flex SQ

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2009-02; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
IgE-blocking factor | start of treatment and 1 week after end of treatment

SECONDARY OUTCOMES:
Tolerability of two different updosing schedules | throughout treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Jung, MD, Principal Investigator — Private practice, Erfurt, Germany
Locations (1):
- Allergists' practice Dr. Kirsten Jung, Erfurt, Thuringia, Germany

REFERENCES:
- [Result] Pfaar O, Jung K, Wolf H, Decot E, Kleine-Tebbe J, Klimek L, Wustenberg E. Immunological effects and tolerability of a new fast updosed immunologically enhanced subcutaneous immunotherapy formulation with optimized allergen/adjuvant ratio. Allergy. 2012 May;67(5):630-7. doi: 10.1111/j.1398-9995.2012.02801.x. Epub 2012 Mar 3. PMID 22385366